CLINICAL TRIAL: NCT03430050
Title: Progesterone for the Treatment of Cannabis Withdrawal
Brief Title: Progesterone for Cannabis Withdrawal
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65954; 5K24DA038240-03 (NIH)
Record Dates: First submitted 2018-01-10; First posted 2018-02-12 (Actual); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Cannabis Use Disorder; Cannabis Withdrawal
Keywords: Progesterone; Ovarian hormones; Gender; Cannabis; Withdrawal; Cognitive functioning
MeSH Terms: conditions — Coitus; Marijuana Abuse | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Progesterone (Active Comparator): Prometrium 200mg. Take one pill in the evening on day 1 with water. Take one pill twice a day on days 2-4. Take one pill on morning day 5.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): Placebo. ake one pill in the evening on day 1 with water. Take one pill twice a day on days 2-4. Take one pill on morning day 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Progesterone capsule
  Other Names: Prometrium
  Arms: Progesterone
Drug: Placebo — Placebo capsule. Manufactured to mimic progesterone 200mg capsule.
  Other Names: Inactive comparator
  Arms: Placebo

SUMMARY:
Sex and gender differences in behavioral, biological, and clinical correlates of substance use disorders are myriad, yet there exists a dearth of gender-informed treatment options. Ovarian hormones have been identified as potential mechanisms of these disparities , and recent clinical trials have begun to examine their utility as possible pharmacotherapeutic agents. The ovarian hormone progesterone has shown promise as a treatment for female cocaine and nicotine users, but has not yet been tested for cannabis. Gender differences in cannabis withdrawal, which is associated with relapse, are pronounced and several studies report more severe and impairing withdrawal symptoms in women compared to men. Developing pharmacological interventions for cannabis withdrawal remains an important priority given the significant cognitive, psychiatric, and physical consequences of heavy cannabis use.

DETAILED DESCRIPTION:
Substantial evidence demonstrates sex and gender differences in the behavioral, biological, and clinical correlates of substance use disorders. Men tend to initiate use earlier and have higher lifetime prevalence rates of disorder, but women demonstrate more severe withdrawal, more rapid progression from first use to disorder, and greater likelihood of comorbid psychiatric disorder. A growing literature suggests that the ovarian hormones progesterone and estradiol may play a key role in these differences. Evidence from preclinical and clinical research suggests that estradiol enhances drug sensitivity and related behavior, while progesterone attenuates drug sensitivity and behavior. As such, recent clinical trials investigating exogenous progesterone as a potential pharmacologic intervention have shown attenuated subjective and physiological effects of cocaine and nicotine in drug-dependent women, and improved cognitive performance in female smokers. While progesterone has shown promise as a treatment for women with cocaine and nicotine use disorder, it has not yet been tested for cannabis.

To date, there are no approved pharmacologic interventions for cannabis use disorder (CUD) despite numerous clinical trials. Cannabis withdrawal is one potential target for CUD medication development research as withdrawal increases risk of relapse. Important gender differences in cannabis withdrawal have been identified warranting gender-based investigation. Several studies have found that women experience more severe and impairing withdrawal symptoms, primarily physiological (e.g. stomach aches, headaches, nausea) and mood-related (e.g. irritability, mood swings), compared to men. As a naturally occurring sex hormone, progesterone may effectively address these gender differences. The proposed pilot study investigates the feasibility and efficacy of exogenous progesterone administration for cannabis withdrawal among female cannabis users.

Specific Aim 1: Test the feasibility of exogenous progesterone administration among cannabis users.

Hypothesis 1: Exogenous progesterone administration will induce normative elevations in progesterone comparable to the luteal phase of female menstrual cycle and will be well-tolerated by participants.

Specific Aim 2: Examine the efficacy of exogenous progesterone on cannabis withdrawal.

Hypothesis 2: Compared to placebo, progesterone will attenuate withdrawal symptoms among heavy-cannabis-using women.

Exploratory Aim: Examine the effect of exogenous progesterone on cognitive functioning during cannabis withdrawal.

Exploratory hypothesis: Compared to placebo, progesterone will enhance cognitive functioning among heavy-cannabis-using women.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments and study procedures.
2. Age 18-45, with regular menses (every 25-35 days).
3. Report using cannabis at least 5 days per week, for at least the past year.
4. Consent to remain abstinent from alcohol for 12 hours prior to study visits, and all other drugs other than cannabis or nicotine for the duration of the study.
5. Consent to random assignment.

Exclusion Criteria:

1. Participants who are pregnant, nursing, amennorheic, or using oral contraceptives.
2. History of major medical illnesses; including liver diseases, abnormal vaginal bleeding, suspected or known malignancy, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke or other medical conditions that the investigator deems as contraindicated for the patient to be in the study;
3. Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent/current psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder.
4. Current suicidal or homicidal risk. Any subject who endorses suicidal ideation will be seen by a licensed clinician in the Addiction Sciences Division who will determine the best course of action to ensure patient safety.
5. Known allergy to progesterone or peanuts (vehicle for micronized progesterone).
6. Unwilling or unable to maintain abstinence from alcohol 12 hours prior to study visits, and all other drugs other than cannabis or nicotine for the duration of the study.
7. Meet DSM-5 criteria for moderate to severe substance use disorder (other than nicotine, cannabis, or alcohol) within the past year.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Normally cycling menstruating females.
Enrollment: 8 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Sherman, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Progesterone | Placebo
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Progesterone Level
Description: Participants took progesterone or placebo for 5 days. Salivary progesterone was measured each day. Change score was calculating by subtracting Day 1 progesterone levels from Day 5 progesterone levels.
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 3 | 5
pg/ml | 237.86 (24.21) | 97.87 (14.67)

2. Primary Outcome: Change in Cannabis Withdrawal Scale Score.
Description: Participants took progesterone or placebo for 5 days. The Cannabis Withdrawal Scale was administered each day. The 19-item scale is used to measure cannabis withdrawal symptoms and negative impact on daily life. The item scores range from 0 - not at all to 10- Extremely. Scores on all items are summed to attain the scale score, so individuals can score between 0-190. Higher scores indicates more severe withdrawal symptoms and greater negative impact. Change score was calculating by subtracting Day 1 CWS scores from Day 5 CWS scores. A positive change score reflects an increase in withdrawal symptoms, while a negative change score reflects a decrease in withdrawal symptoms.
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 3 | 5
units on a scale | 29.08 (4.15) | 20.41 (3.18)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Progesterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03430050/Prot_SAP_000.pdf